CLINICAL TRIAL: NCT06682403
Title: Hospital Security Program for Engaging Communities With Firearm Safe Storage Devices and Interventions
Brief Title: Distribution and Randomization of Gun Safety Devices to Measure Uptake and Preferences
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, M. Kit Delgado, MD, Associate Professor of Emergency Medicine and Epidemiology, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 855259
Record Dates: First submitted 2024-06-07; First posted 2024-11-12 (Actual); Results first posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Gun Violence Prevention

STUDY DESIGN:
Intervention Model Description: Participants who fill out the survey linked to study posters and brochures will be randomized to either receive a cable lock as the default safety device option or the choice between a cable lock or lock box, shipped to their address. For individuals who take a cable lock at time of receiving a brochure, they are automatically assigned into the cable lock group.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individual receives cable lock as default (Experimental): Participants in this arm are either automatically assigned due to taking a cable lock at the hospital when offered AND fill out the survey OR are randomized into this group by filling out the study survey linked in study materials.
  Interventions: Behavioral: Received cable lock as default
- Individual has a choice between cable lock and lock box (Experimental): Participants in this arm are randomized into it based on NOT taking a cable lock at the hospital when offered AND fill out the survey OR are randomized into this group by filling out the study survey linked in study materials.
  Interventions: Behavioral: Choice between cable lock or lock box

INTERVENTIONS:
Behavioral: Received cable lock as default — Participants will receive a cable lock as the default safety device option after filling out the survey. If the participant took a cable lock during their hospital visit and noted this in the survey, they will not be shipped a cable lock. If participants did not take a cable lock and noted this in the survey, they will be shipped a cable lock.
  Arms: Individual receives cable lock as default
Behavioral: Choice between cable lock or lock box — Participant will have the option to select a lock box or cable lock shipped to their address after filling out the study survey.
  Arms: Individual has a choice between cable lock and lock box

SUMMARY:
This study aims to enhance workplace safety by implementing a firearm safety program at Penn Medicine Pennsylvania Hospital (PAH). The option to store firearms securely during visits is offered to firearm owners. The study focuses on understanding barriers and facilitators to this program and piloting methods to collect data on firearm storage device use. The approach prioritizes participant confidentiality and pragmatism. The study design involves iterative pilot testing of data collection methods and comparison of acceptance and usage rates between cable locks and lock boxes through randomization. The intended outcome is to provide evidence supporting the scalability and effectiveness of the program. The study population includes patients and visitors who accept firearm safety materials or express interest in receiving a firearm storage device. The primary outcome measure is survey response rate, with secondary outcomes including firearm storage behavior and likelihood of using a gun safety device. Additionally, the study explores variations in survey distribution methods.

DETAILED DESCRIPTION:
To prevent workplace violence, in November 2021, Penn Medicine implemented the Evolv weapons detection system in Pennsylvania Hospital (PAH) (1,2). For individuals who self-disclose they are carrying a weapon, or who are identified with weapon during screening, security guards offer the individual the option to leave with weapon, or to place it in a safe, at the hospital, for storage. Security guards return the weapon when the patient or visitor is ready to leave. Beginning in July 2022 team piloted a program in which security guards offer a cable lock and safety brochure when the gun owner returns to retrieve firearm at the conclusion of visit. To date, 47% of patients and visitors who stored a firearm with security have taken a cable lock when offered, resulting in over 400 firearm safety locks and brochures distributed to firearm owners. The Aims of this study are to: (1) Elucidate barriers and facilitators to implementing a hospital security screening firearm safety program through interviews with hospital security staff; (2) Design and pilot test a method for collecting data on storage device use among patients and visitors who accept firearm safety materials; (3) Conduct a pilot of distributing lockboxes and compare acceptance and usage rates to cable locks.

This protocol is for Aim 2 and 3 of the study. The rationale for this aim is that traditional research methods for collecting data on firearm safe storage have not been optimized for use in a pragmatic setting to ensure acceptability and confidentiality. Priority in firearm safety education and device distribution is to get the necessary information and supplies to those in need or desire such resources. To achieve this, any data collection must be done in a low profile, confidential, and non-threatening way. This is particularly important not only because discussions of firearm ownership can be politically charged, but also because some community members may not be legally licensed to own or carry a firearm, and some may even be legally prohibited from doing so. The legal status of gun ownership does not lessen the need for safety information and support-indeed, unlicensed firearm owners may have even fewer safety resources available for the. Priority is therefore to reach as many individuals as possible while subjecting participants to as little scrutiny as possible. Therefore, the aim is to design a data collection approach that will prioritize preserving participant confidentiality. Approach will be iterative pilot tests of data collection methods including embedding unique quick response (QR) codes linked to surveys in firearm safety brochures and study poster signage. The opportunity will be offered for individuals to take home a cable lock after visiting or to scan the QR code on the brochure/poster to fill out the study survey and get a safety device shipped to a participant address. Participants who fill out the study survey will be randomized to receive either a cable lock as the default or a choice between cable lock and lock box to test acceptance and usage rates. For those who accepted a cable lock at the hospital will automatically be grouped in the cable lock default group. The hypothesis that is being tested is if iterative pilot testing will reveal a feasible method that balances pragmatism and confidentiality as well as compare acceptance and usage rates among cable locks and lock boxes.

The intended outcome of this study is development of critical evidence to facilitate the scaling of this program to other hospitals and launch a promising research program to study the acceptability, long term use, and cost-effectiveness of a scalable approach to promote safe firearm storage.

This research study is to design and pilot test a method for collecting data on storage device use among patients and visitors who accept firearm safety materials or are interested in receiving a firearm storage device shipped to the participant's address. The study design is an iterative pilot test of survey data collection methods and determination of scalability and feasibility for distribution of firearm storage devices. The study population and sample will be (a) individuals who are patients or visitors to PAH who are screened for a firearm, screen positive, and accept a firearm safety brochure and storage device OR (b) individuals interested in receiving a firearm storage device and self-scan the unique QR code on the study poster in the entry hall of PAH with minimal or no security supervisor engagement. A unique QR code linking directly to the initial survey will be embedded into the firearm safety brochure as well as the poster in the entry hall of PAH next to the distribution area. Individual group (a) will be informed by security that survey participation is optional, but that it is helpful for efforts. Individual group (b) will not be actively engaged by security, and will self-enroll in the study by viewing the posted signage and completing the QR code linked survey.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals who are visitors or patients at Penn Medicine Facilitates who are identified through security screening as carrying a firearm, and who accept a firearm safety brochure and scan the QR code in the brochure; OR
2. Any patient or visitor interested in receiving a firearm storage device who self-selects into the study by scanning the QR code on the study poster; OR
3. Any individual interested in receiving a firearm storage device who clicks the link to the survey posted on the Penn Medicine Safety Measures website that is included health system appointment reminders.

Exclusion Criteria:

* Individuals who have already completed the survey or have already requested a gun safety device.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mucio K Delgado, MD, Principal Investigator — University of Pennsylvania; Elinore Kaufman, MD, Principal Investigator — University of Pennsylvania; Katelin Hoskins, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Pennsylvania Hospital, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Cunningham RM, Walton MA, Carter PM. The Major Causes of Death in Children and Adolescents in the United States. N Engl J Med. 2018 Dec 20;379(25):2468-2475. doi: 10.1056/NEJMsr1804754. No abstract available. PMID 30575483
- See also: Patient charged in stabbing of doctor at Pennsylvania Hospital — https://www.inquirer.com/news/penn-medicine-pennsylvania-hospital-doctor-stabbed-violence-police-arrest-philadelphia-20210223.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Individual Receives Cable Lock as Default | Individual Has a Choice Between Cable Lock and Lock Box
Started | 25 | 24
Completed | 25 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: A total of 45 participants who reported having firearms at home were enrolled and randomized equally into two arms: one group received cable locks, and the other was given a choice between a cable lock or a lockbox. All baseline data were collected via a voluntary, anonymous online survey completed at enrollment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Individual Receives Cable Lock as Default | Individual Has a Choice Between Cable Lock and Lock Box | Total
Number analyzed (Participants) | 23 | 22 | 45
Age, Categorical [Count of Participants; unit: Participants] — Population: Age data were not collected as part of the anonymous survey.
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Sex (Female, Male) were not collected due to the anonymous nature of the survey.
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23 | 22 | 45
Visited Pennsylvania Hospital during the study period [Count of Participants; unit: Participants] | 23 | 22 | 45

OUTCOME MEASURES:

1. Primary Outcome: Survey Response Rate
Description: The primary outcome measure is survey response rate, defined as whether an eligible visitor or patient completed the firearm storage survey after accepting firearm safety materials or after scanning the QR code on the study poster.
Time Frame: From 2 to 4 weeks
Population: All participants included in the analysis were patients or visitors at Pennsylvania Hospital who self-enrolled via QR code from study signage. Participants were grouped into two arms: those who received only a cable lock and those offered a choice between a cable lock and a lockbox. Survey response rates were analyzed at baseline, 2-week, and 4-week time points.
Measure: Count of Participants; unit: Participants
Groups:
- Baseline: Initial survey administered upon firearm safety device offer or QR scan from brochure/poster.
- Follow-up #1 (2-week): First follow-up survey sent via text two weeks post-enrollment.
- Follow-up #2 (4-week): Second optional follow-up survey at 4 weeks for continued behavior tracking.
Arm/Group | Baseline | Follow-up #1 (2-week) | Follow-up #2 (4-week)
Number analyzed (Participants) | 45 | 45 | 45
Participants
  Respond (Yes): number analyzed (Participants) | 45 | 28 | 24
  Respond (Yes): Cable Lock Only Group | 23 | 15 | 14
  Respond (Yes): Choice of Lock Group | 22 | 13 | 10
  Respond (No): number analyzed (Participants) | 0 | 17 | 21
  Respond (No): Cable Lock Only Group | 0 | 8 | 9
  Respond (No): Choice of Lock Group | 0 | 9 | 12

2. Secondary Outcome: Rate of Full Firearm Storage at Follow-Up
Description: The secondary outcome was the rate of full firearm storage, defined as participants who responded "Yes, all of them" on the follow-up survey. Of the 45 participants who reported having a firearm at home and received the safety devices, 28 completed the first follow-up survey and were included in the primary outcome analysis. Among the 28 participants who completed the first follow-up, 24 responded to the second follow-up survey. 17 participants did not respond to the first follow-up survey and were therefore excluded from the analysis.
Time Frame: From 2 to 4 weeks
Population: Participants who completed the follow-up survey and reported having a firearm at home.
Measure: Count of Participants; unit: Participants
Arm/Group | Individual Receives Cable Lock as Default | Individual Has a Choice Between Cable Lock and Lock Box
Number analyzed (Participants) | 15 | 13
Participants
  First Follow-Up | 13 | 11
  Second Follow-Up: number analyzed (Participants) | 14 | 10
  Second Follow-Up | 12 | 7

3. Secondary Outcome: Likelihood of Using Cable Lock Within the Next Week (Extremely Unlikely to Extremely Likely Scale).
Description: The survey were asked to indicate their likelihood of using the device within the next week. Responses were collected using a 5-point Likert scale ranging from "Extremely unlikely" to "Extremely likely." This measure is intended to assess anticipated short-term behavior change related to firearm safe storage following receipt of a safety device. Responses are collected through an initial Qualtrics web-based survey and analyzed as part of the study's secondary outcomes to evaluate the acceptability and intended use of the distributed firearm safety materials.
Time Frame: From 2 to 4 weeks
Population: This analysis includes participants who accepted a cable lock and completed the initial Qualtrics survey by scanning the QR code from the study poster. A total of 45 participants responded to the question regarding their likelihood of using the cable lock within the next week. Responses with missing data for this question (n=5) were counted as "Missing" in the data table.
Measure: Count of Participants; unit: Participants
Groups:
- How Likely Are You to Use Your New Cable Lock in the Next Week?, n (%): Participants who completed the initial survey by scanning the study poster QR code. In the Qualtrics Survey, individuals were asked how likely they were to use the cable lock within the next week.
Arm/Group | How Likely Are You to Use Your New Cable Lock in the Next Week?, n (%)
Number analyzed (Participants) | 45
Participants
  Very likely | 37
  Somewhat likely | 2
  Neither likely nor unlikely | 1
  Somewhat unlikely | 0
  Very unlikely | 0
  Missing | 5

ADVERSE EVENTS:
Description: No adverse event data were collected for this study. Adverse event monitoring was not part of the study design.
Arm/Group | Individual Receives Cable Lock as Default | Individual Has a Choice Between Cable Lock and Lock Box
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-01-16): https://cdn.clinicaltrials.gov/large-docs/03/NCT06682403/Prot_000.pdf
  • Informed Consent Form (2024-01-16): https://cdn.clinicaltrials.gov/large-docs/03/NCT06682403/ICF_001.pdf